CLINICAL TRIAL: NCT04323514
Title: Use of Ascorbic Acid in Patients With COVID 19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Salvatore Corrao, MD, Professor, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3143
Record Dates: First submitted 2020-03-18; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Hospitalized Patients With Covid-19 Pneumonia
Keywords: pneumonia; covid-19; hospitalized patients; vitamin C
MeSH Terms: conditions — Pneumonia; COVID-19 | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with COVID-19 pneumonia (Experimental): Consecutive patients with COVID-19 pneumonia admitted to ARNAS Civico-Di Cristina-Benfratelli, Palermo
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — 10 gr of vitamin C intravenously in addition to conventional therapy.

SUMMARY:
Different studies showed that ascorbic acid (vitaminC) positively affects the development and maturation of T-lymphocytes, in particular NK (natural Killer) cells involved in the immune response to viral agents. It also contributes to the inhibition of ROS production and to the remodulation of the cytokine network typical of systemic inflammatory syndrome.

Recent studies have also demonstrated the effectiveness of vitamin C administration in terms of reducing mortality, in patients with sepsis hospitalized in intensive care wards.

Given this background, in the light of the current COVID-19 emergency, since the investigators cannot carry out a randomized controlled trial, it is their intention to conduct a study in the cohort of hospitalized patients with covid-19 pneumonia, administering 10 gr of vitamin C intravenously in addition to conventional therapy.

DETAILED DESCRIPTION:
The Sars-COV-2, has spread all over the world, in two months after its discovery in China. Outbreaks have been reported in more than 50 countries with more than 118,223 confirmed cases and 4,291 deaths worldwide. In Italy, the scenario is progressively worsening with 8514 confirmed cases and 631 deaths at 10/3/2020.

Along with the spread of this new virus there has been an increase in the number of pneumonia identified with the term novel coronavirus (2019-nCoV)-infected pneumonia (NCIP), which are characterized by fever, asthenia, dry cough, lymphopenia, prolonged prothrombin time, elevated lactic dehydrogenase, and a tomographic imaging indicative of interstitial pneumonia (ground glass and patchy shadows).

Recent studies have shown the efficacy of vitamin C and thiamine administration in patients hospitalized for sepsis in the setting of intensive wards in terms of mortality reduction. The use of intravenously vitamin C arises from the experimental evidence of its anti-inflammatory and antioxidant properties. Vitamin C causes a greater proliferation of natural killers without affecting their functionality. Moreover, the vitamin C reduces the production of ROS (reactive oxygen species) that contribute to the activation of the inflammosomi and, in particular, the NLRP3 that affetcs the maturation and secretion of cytokines such as IL1beta and IL-18 that are involved in the inflammatory systemic syndrome that characterized sepsis. Vitamin C blocks the expression of ICAM-1 and activation of NFKappaB that are involved in inflammatory, neoplastic, and apoptotic processes by the inhibition of TNFalfa.

For this reason, the use of vitamin C could be effective in terms of mortality and secondary outcomes in the cohort of patients with covid-19 pneumonia.

In view of the emergency of SARS-VOC-2 and the impossibility of carrying out a randomized controlled study, it is their intention to conduct an intervention protocol (administration of 10 grams of vitamin C intravenously in addition to conventional therapy) involving the cohort of hospitalized patients with covid-19 pneumonia.

Methods:

An uncontrolled longitudinal study will be conducted at the Arnas Civico-di Cristina-Benfratelli National Relevance Hospital in Palermo. This study will include all patients consecutively hospitalized with positive swab test of SARS-CoV-2 and interstitial pneumonia or with interstitial pneumonia with indication of intubation. At the admission, data will be collected: personal and anamnestic information, clinical and laboratory findings such as Gender, Age, Ethnicity, Comorbidities, Drugs, blood urea nitrogen, Creatinine, Electrolytes, Blood cell count, Clearance of the lactates, PCR, PCT, SOFA score, liver function, Coagulation, Blood gas analysis, Systolic and Diastolic Blood Pressure, Sp02, Glycaemia, Body Mass Index (BMI). Length of hospital stay will be recorded. After written informed consent, 10 grams of vitamin C in 250 ml of saline to infuse at a rate of 60 drops / minute will be administered. In-hospital mortality, reduction of PCR levels > 50% in comparison with PCR levels at the admission within 72 hours after the administration, lactate clearance, length of hospital stay, resolution of symptoms, duration of positive swab (days). Resolution of the CT imaging will be analysed. Stata Statistical Software: Release 14.1. College Station, TX: StataCorp LP) was used for database management and analysis.

ELIGIBILITY:
Inclusion Criteria:

* In case of doubt of interstitial pneumonia with indications for intubation
* Positive swab test of SARS-CoV-2
* Interstitial pneumonia
* Signature of informed consent

Exclusion Criteria:

* Unsigned informed consent
* Negative swab test of SARS-CoV-2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-03-13 (Estimated); Study Completion 2021-03-13 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 72 hours
  Change of hospital mortality

SECONDARY OUTCOMES:
PCR levels | 72 hours
  Reduction of PCR levels > 50% in comparison with PCR levels at the admission, within 72 hours after the administration
Lactate clearance | 72 hours
  Change of the lactate clearance
Hospital stay | 72 hours
  Change of hospital stay days
Symptoms | 72 hours
  Resolution of symptoms (Fever, Cough, Shortness of breath or difficulty breathing)
Positive swab | 72 hours
  Change of duration of positive swab (nasopharynx and throat)
Tomography imaging | 72 hours
  Resolution of tomography imaging (example, patches located in the subpleural regions of the lung)

CONTACTS AND LOCATIONS:
Locations (1):
- A.R.N.A.S. Civico - Di Cristina - Benfratelli, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT04323514/Prot_SAP_ICF_000.pdf